CLINICAL TRIAL: NCT03235804
Title: The Impact of a Powdered Meal Replacement on Metabolism and Gut Microbiota: a 12-week Study in Individuals With Excessive Body Weight
Brief Title: The Impact of a Powdered Meal Replacement on Metabolism and Gut Microbiota
Acronym: PREMIUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Almased Wellness GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00070712
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Dietary Modification
Keywords: Powdered meal replacement; Inflammation; Gut microbiota; Energy metabolism; Body composition
MeSH Terms: conditions — Inflammation | interventions — Soybean Proteins; Honey; Yogurt

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Those assigned to the Control group will be asked to maintain their usual dietary intake over 12 weeks. Participants' usual dietary intake is expected to reflect the North American dietary pattern (i.e. ~15% of total energy intake coming from protein, ~50% from carbohydrate and ~35% from fat).
- Powdered Meal Replacement Group (Experimental): Those assigned to the Powdered Meal Replacement group will be asked to maintain their usual dietary intake and consume a powdered meal replacement composed of soy protein, honey and yogurt twice daily (in two snacks) over 12 weeks. The addition of the nutritional supplement to a North American Dietary Pattern (described on the CON group diet) will result in a diet composed of, approximately, 22% of protein, 48% of carbohydrate and 30% of fat of total energy intake. The amount of protein is considered higher than the North American dietary pattern (i.e. 15%); however, still within the Acceptable Macronutrient Distribution Range (AMDR) recommended by the Dietary Guidelines for Americans (10-35%).
  Interventions: Dietary Supplement: Soy protein, honey and yogurt.

INTERVENTIONS:
Dietary Supplement: Soy protein, honey and yogurt. — Participants will be asked to maintain their usual dietary intake and consume a powdered meal replacement composed of soy protein, honey and yogurt twice daily (in two snacks) over 12 weeks. The addition of the nutritional supplement to a North American Dietary Pattern (described on the CON group diet) will result in a diet composed of, approximately, 22% of protein, 48% of carbohydrate and 30% of fat of total energy intake. The amount of protein is considered higher than the North American dietary pattern (i.e. 15%); however, still within the Acceptable Macronutrient Distribution Range (AMDR) recommended by the Dietary Guidelines for Americans (10-35%).
  Arms: Powdered Meal Replacement Group

SUMMARY:
This study will investigate the impact of a 12-week powdered meal replacement on inflammatory, metabolic, and hormonal markers of obesity-associated conditions and to correlate this response to compositional shifts within the gut microbiota. Moreover, resting energy expenditure, body composition, appetite sensations and soy metabolomics will be explored.

This study will be a randomized, parallel group, clinical trial of a 12-week nutritional intervention. A sample size of n=88 participants will be randomly allocated into one of the following groups:

* Control group (CON): Participants will be asked to maintain their usual dietary intake over 12 weeks. Their usual dietary intake is expected to reflect the North American dietary pattern (i.e. ~15% of total energy intake coming from protein, ~50% from carbohydrate and ~35% from fat).
* Powdered Meal Replacement group (PMR): Participants will be asked to maintain their usual dietary intake and consume a powdered meal replacement composed of soy protein, honey and yogurt twice daily (in two snacks) over 12 weeks. The addition of the meal replacement to a North American Dietary Pattern (described on the CON group diet) will result in a diet composed of, approximately, 22% of protein, 48% of carbohydrate and 30% of fat of total energy intake.

The following variables will be analyzed:

* Interleukin (IL)-6.
* Gut microbiota diversity and composition, specifically taxa that have been associated with health benefits, obesity, and weight loss.
* Systemic inflammatory biomarkers (high-sensitivity C-reactive protein, IL-8, IL-10 and tumor necrosis factor-α);
* Metabolic blood markers (glucose, insulin, lipid panel, peptide tyrosine-tyrosine, glucagon-like peptide-1, ghrelin, adiponectin, leptin, free glycerol, free fatty acids, and thyroid stimulating hormone)
* Resting energy expenditure;
* Body composition;
* Appetite sensations (hunger, satiety, fullness, and prospective food consumption);
* Soy polyphenols' metabolomics.
* Gene expression and genetic polymorphisms. At baseline and after 6 and 12 weeks, individuals will attend our Human Nutrition Research Unit where all assessments will take place. In order to assess participants' adherence and follow-up, dietary intake, body weight and appetite sensations (only for participants assigned to the PMR group) will be assessed weekly during the 12-week intervention period. Additionally, participants will be contacted by phone weekly and reminded to maintain their journal/log.

DETAILED DESCRIPTION:
Overweight and obesity increase the risk of developing several diseases having a negative effect on people's health. The prevalence of these conditions is increasing worldwide, but successful treatments are lacking. As excess body weight is a result of an imbalance between calories in and calories out, dietary intake plays an important role in maintaining a healthy body weight and overall health status. Meal replacements are nutritionally complete formula foods used to substitute a meal. They can be a drink, bar, or soup. These products have been gaining popularity because they can help individuals lose weight. In addition, depending on its ingredients, meal replacements may affect our health. For this reason, meal replacements have been studied for health benefits. However, how meal replacements affect the microbes living in our gut, inflammation, and our genes is not known. Well-designed studies using state-of-the-art equipment can help elucidate the mechanisms by meal replacements act in individuals with overweight or obesity.

The overall purpose of this research is to investigate the impact of a 12-week powdered meal replacement on inflammatory, metabolic, and hormonal markers of obesity-associated conditions and to correlate this response to compositional shifts within the gut microbiota. Moreover, resting energy expenditure, body composition, appetite sensations, soy metabolomics, gene expression, and genetic polymorphisms will be explored.

This study will be a randomized, parallel group, clinical trial of a 12-week nutritional intervention. A sample size of n=88 participants will be randomly allocated into one of the following groups:

* Control group (CON): Participants will be asked to maintain their usual dietary intake over 12 weeks. Participants' usual dietary intake is expected to reflect the North American dietary pattern (i.e. ~15% of total energy intake coming from protein, ~50% from carbohydrate and ~35% from fat).
* Powdered Meal Replacement group (PMR): Participants will be asked to maintain their usual dietary intake and consume a powdered meal replacement composed of soy protein, honey and yogurt twice daily (in two snacks) over 12 weeks. The addition of the nutritional supplement to a North American Dietary Pattern (described on the CON group diet) will result in a diet composed of, approximately, 22% of protein, 48% of carbohydrate and 30% of fat of total energy intake. The amount of protein is considered higher than the North American dietary pattern (i.e. 15%); however, still within the Acceptable Macronutrient Distribution Range (AMDR) recommended by the Dietary Guidelines for Americans (10-35%).

The following variables will be analyzed:

* Interleukin (IL)-6.
* Gut microbiota diversity and composition, specifically taxa that have been associated with health benefits, obesity, and weight loss.
* Systemic inflammatory biomarkers (high-sensitivity C-reactive protein [hs-CRP], IL-8, IL-10 and tumor necrosis factor-α [TNF-α]);
* Metabolic blood markers [glucose, insulin, lipid panel (i.e. total cholesterol, LDL, HDL, and triglycerides), peptide tyrosine-tyrosine (PYY), glucagon-like peptide-1 (GLP-1), ghrelin, adiponectin, leptin, free glycerol, free fatty acids, and thyroid stimulating hormone (TSH)];
* Resting energy expenditure;
* Body composition;
* Appetite sensations (hunger, satiety, fullness, and prospective food consumption);
* Soy polyphenols' metabolomics.
* Gene expression and genetic polymorphisms. At baseline and after 6 and 12 weeks, individuals will attend our Human Nutrition Research Unit where all assessments will take place. In order to assess participants' adherence and follow-up, dietary intake, body weight and appetite sensations will be assessed weekly during the 12-week intervention period. Additionally, participants will be contacted by phone weekly and reminded to maintain their journal/log. Dietary intake will be assessed by a 3-day dietary record (2 week days and 1 weekend day) at baseline, at mid-point and end of the study. Participants will also be asked to complete a 1-day dietary record on one weekday, each week of the study. The purpose of this regular assessment is to avoid daily fluctuations in eating patterns, also ensuring a personalized feedback for those experiencing weight fluctuations. Both of these assessments (i.e. 1-day and 3-day dietary records) will be conducted using the online Automated Self -Administered 24-hour Recall (ASA24) Canada. The ASA24 is a validated web-based program that uses the validated U.S. Department of Agriculture's Automated Multiple-Pass Method, and is modified to support the Canadian food supply.

Participants will receive a digital scale and will be asked to weight themselves daily. Participants from the PMR group will also be asked to rate their appetite sensations on a 100-mm VAS paper sheet. Appetite sensation should be completed in the morning (after waking up and while fasting) and 30 minutes after consuming the supplement snacks in order to assess hunger, satiety, fullness, and prospective food consumption.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker;
* Female/Male;
* Aged 18 to 50 years;
* Body mass index (BMI) between 25 and 37 kg/m²;
* Weight stable (< ± 5 kg over past 6 months);
* Fat mass ≥20% for men and ≥25% for women;
* Maintaining current levels of physical activity throughout the study.
* Female participants must verify use of acceptable, effective birth control methods (total abstinence, hormonal birth control [oral, injectable, transdermal, intravaginal], intrauterine devices, confirmed successful vasectomy or partner, or condoms).

Exclusion Criteria:

* Diagnosis of chronic diseases or acute infections;
* Taking any medication that may alter inflammation, energy metabolism, body weight and composition, gut microbiota and hormone levels; investigators should always be informed if there are any changes in medications or Natural health product use;
* Taking pre- and probiotics (e.g. supplements);
* Use of antibiotics in the past two months;
* Use of thyroid replacement therapy;
* Use of nutritional supplements in the past four weeks (multivitamin and vitamin D3 are permitted to be used during the course of the study);
* Allergy to any ingredient (including non-medicinal ingredients) in investigational product;
* Lactose, gluten and/or soy allergic/intolerant;
* Follow a vegetarian, vegan or any restrictive dietary pattern;
* Pregnant or lactating;
* Perform over three hours of vigorous physical activity per week;
* A nuclear medicine scan or injection of an X-ray dye in the past week;
* A barium test/exam in the last two weeks;
* Suffer from claustrophobia;
* Inability to comprehend and complete the required questionnaires.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Interleukin-6. | At baseline (week 1), middle (week 6) and end (week 12) of the intervention period (12 weeks).
  Changes in blood interleukin-6 will be assessed at baseline, middle and end of the 12-week dietary intervention period.

SECONDARY OUTCOMES:
Gut microbiota diversity and composition. | At baseline (week 1), middle (week 6) and end (week 12) of the intervention period (12 weeks).
  Changes in gut microbiome diversity and composition (specifically taxa that have been associated with health benefits, obesity and weight loss) will be assessed at baseline, middle and end of the 12-week dietary intervention period.

OTHER OUTCOMES:
High-sensitivity C-reactive protein. | At baseline (week 1), middle (week 6) and end (week 12) of the intervention period (12 weeks).
  Changes in blood high-sensitivity C-reactive protein will be assessed at baseline, middle and end of the 12-week dietary intervention period.
Interleukin 8. | At baseline (week 1), middle (week 6) and end (week 12) of the intervention period (12 weeks).
  Changes in interleukin 8 will be assessed at baseline, middle and end of the 12-week dietary intervention period.
Interleukin 10. | At baseline (week 1), middle (week 6) and end (week 12) of the intervention period (12 weeks).
  Changes in interleukin 10 will be assessed at baseline, middle and end of the 12-week dietary intervention period.
Tumor necrosis factor-α. | At baseline (week 1), middle (week 6) and end (week 12) of the intervention period (12 weeks).
  Changes in tumor necrosis factor-α will be assessed at baseline, middle and end of the 12-week dietary intervention period.
Adiponectin. | At baseline (week 1), middle (week 6) and end (week 12) of the intervention period (12 weeks).
  Changes in adiponectin will be assessed at baseline, middle and end of the 12-week dietary intervention period.
Blood glucose. | At baseline (week 1), middle (week 6) and end (week 12) of the intervention period (12 weeks).
  Changes in blood glucose will be assessed at baseline, middle and end of the 12-week dietary intervention period.
Insulin. | At baseline (week 1), middle (week 6) and end (week 12) of the intervention period (12 weeks).
  Changes in insulin will be assessed at baseline, middle and end of the 12-week dietary intervention period.
Lipid panel. | At baseline (week 1), middle (week 6) and end (week 12) of the intervention period (12 weeks).
  Changes in lipid panel (i.e. total cholesterol, LDL, HDL and triglycerides) will be assessed at baseline, middle and end of the 12-week dietary intervention period.
Peptide tyrosine-tyrosine. | At baseline (week 1), middle (week 6) and end (week 12) of the intervention period (12 weeks).
  Changes in peptide tyrosine-tyrosine will be assessed at baseline, middle and end of the 12-week dietary intervention period.
Glucagon-like peptide 1. | At baseline (week 1), middle (week 6) and end (week 12) of the intervention period (12 weeks).
  Changes in glucagon-like peptide-1 will be assessed at baseline, middle and end of the 12-week dietary intervention period.
Ghrelin. | At baseline (week 1), middle (week 6) and end (week 12) of the intervention period (12 weeks).
  Changes in ghrelin will be assessed at baseline, middle and end of the 12-week dietary intervention period.
Leptin. | At baseline (week 1), middle (week 6) and end (week 12) of the intervention period (12 weeks).
  Changes in leptin will be assessed at baseline, middle and end of the 12-week dietary intervention period.
Free glycerol. | At baseline (week 1), middle (week 6) and end (week 12) of the intervention period (12 weeks).
  Changes free glycerol will be assessed at baseline, middle and end of the 12-week dietary intervention period.
Free fatty acids. | At baseline (week 1), middle (week 6) and end (week 12) of the intervention period (12 weeks).
  Changes in free fatty acids will be assessed at baseline, middle and end of the 12-week dietary intervention period.
Thyroid stimulating hormone. | At baseline (week 1), middle (week 6) and end (week 12) of the intervention period (12 weeks).
  Changes in thyroid stimulating hormone will be assessed at baseline, middle and end of the 12-week dietary intervention period.
Resting energy expenditure. | At baseline (week 1), middle (week 6) and end (week 12) of the intervention period (12 weeks).
  Changes in resting energy expenditure will be assessed at baseline, middle and end of the 12-week dietary intervention period using a whole body calorimetry unit.
Body composition. | At baseline (week 1), middle (week 6) and end (week 12) of the intervention period (12 weeks).
  Changes in fat mass, lean soft tissue and bone mineral content will be assessed at baseline, middle and end of the 12-week dietary intervention period using dual-energy X-ray absorptiometry.
Appetite sensations. | Once per week during the intervention period (12 weeks).
  Changes in hunger, satiety, fullness, and prospective food consumption will be assessed weekly using a 100 mm visual analogue scale.
Soy polyphenols' metabolomics. | At baseline (week 1), middle (week 6) and end (week 12) of the intervention period (12 weeks).
  Soy polyphenols' metabolomics will be assessed on participants assigned to the 12-week dietary intervention periodPowdered Meal Replacement group at baseline, middle and end of the 12-week dietary intervention period using blood and urine samples.
Gene expression | At baseline (week 1) and end (week 12) of the intervention period (12 weeks).
  Changes in gene expression will be assessed at baseline and at the end of the 12-week dietary intervention period
Genetic polymorphisms | At baseline (week 1)
  Genetic polymorphisms will be identified at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jens Walter, PhD, Principal Investigator — University of Alberta; Carla M Prado, PhD, Principal Investigator — University of Alberta; Arya Sharma, PhD, Principal Investigator — University of Alberta
Locations (1):
- Human Nutrition Research Unit, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Montenegro J, L P Oliveira C, Armet AM, Berg A, Sharma AM, Mereu L, Cominetti C, Ghosh S, Richard C, Nguyen NK, Cani PD, Walter J, Prado CM. Impact of a Powdered Meal Replacement on Metabolism and Gut Microbiota (PREMIUM) in individuals with excessive body weight: a study protocol for a randomised controlled trial. BMJ Open. 2023 Sep 13;13(9):e070027. doi: 10.1136/bmjopen-2022-070027. PMID 37709337